CLINICAL TRIAL: NCT06093906
Title: Treatment of Stress-Related Psychopathology: Targeting Maladaptive and Adaptive Event Processing
Brief Title: Positive Processes and Transition to Health (PATH)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University of Washington (Other); University of Delaware (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Norah Feeny, Director, PTSD Treatment and Research Program, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20191519; 4R33MH118401-03 (NIH)
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Posttraumatic Stress Disorder; Major Depressive Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: Participants are randomized to receive PATH therapy or PMR.
Who Masked: Outcomes Assessor
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Processes and Transition to Health (PATH) (Experimental): PATH includes six 60-90 min, weekly sessions, with two booster sessions for partial responders. Session 1 provides the PATH rationale and a review of life events (PATH of life: negative and positive). A rationale for an explicit focus on positive events/emotions will be provided. Sessions 2-4 focus on a verbal narrative of the destabilizing life event, reminiscence and processing of a major positive life event, and real-life practice to enact what was taught. Sessions 5 focuses on constructive processing and provides opportunity for integration and consolidation of learning. Session 6 focuses on future negative and positive events to promote application of new learning and resilience. Booster sessions focus on positive and negative life events since the last session and adaptive processes (constructive processing, approach, and reward). All sessions will include cultivation and elaboration of positive emotions to promote engagement and to build on the benefits of positive emotions.
  Interventions: Behavioral: Positive Processes and Transition to Health
- Progressive Muscle Relaxation (PMR) (Active Comparator): PMR will be adapted from Berstein, Borkoveck, and Hazlett- Stevens (2000). PMR will be conducted in six, 60-90 min individual weekly sessions with a study therapist. Muscle groups are tightened and then relaxed with the attention of the patient focused on the contrast between tension and relaxation. Through regular practice, the person becomes more aware of tension in the body and can induce relaxation as needed (Field, 2009). During the six sessions of training, patients will be encouraged to practice PMR and learn how to deliberately induce physical relaxation to reduce stress and mental tension. Sessions will move from relaxation of 16-muscle groups to 7 muscle groups, 4 muscle groups, and finally to relaxation by recall. Patients will be instructed to practice daily, if possible, but at least two or three times a week, and to integrate the practice into their daily life. They will be provided with audio recordings and homework reporting forms to assist their home PMR exercises.
  Interventions: Behavioral: Progressive Muscle Relaxation

INTERVENTIONS:
Behavioral: Positive Processes and Transition to Health — See arm/group description for details regarding this intervention
  Other Names: PATH
  Arms: Positive Processes and Transition to Health (PATH)
Behavioral: Progressive Muscle Relaxation — See arm/group description for details regarding this intervention
  Other Names: PMR
  Arms: Progressive Muscle Relaxation (PMR)

SUMMARY:
The R33 will be a randomized controlled trial to replicate changes in the targets (unproductive processing, avoidance, reward deficits) from the R61 phase in a larger sample of 135 participants who have experienced a destabilizing life event involving profound loss or threat, report persistent stressor-related symptoms of PTSD and/or depression, and are elevated on symptoms related to 2 of the 3 therapeutic targets. Additionally, this study will examine Positive Processes and Transition to Health (PATH)'s impact on stressor-related psychopathology in comparison to Progressive Muscle Relaxation (PMR). In the R33 phase, the investigators will examine changes in target mechanisms predicting improvements in PTSD and depressive symptoms, as well as feasibility and acceptability. Patients will receive 6 sessions of PATH or PMR (with 2 boosters, if partial responders). Primary targets will be assessed at pre-treatment, week 3, post-treatment, and at 1- and 3-month follow-up; secondary targets at pre-treatment, weekly during treatment, post-treatment, and at 1- and 3-month follow-ups.

DETAILED DESCRIPTION:
Evidence-based psychotherapies for posttraumatic stress disorder (PTSD) and depression consistently produce strong, clinically meaningful effects for many individuals. However, these interventions also have significant dropout rates, a large minority of individuals continue to have debilitating symptoms, and even those who respond may be vulnerable to relapse upon future stressors. More efficient and mechanistically precise interventions are needed. Consistent with the cross-cutting theme of studying the role of the environment in the NIMH Strategic Plan, the etiological role of exposure to destabilizing, stressful life events is common to both PTSD and depression. Not only do they share common distress-related triggers, symptoms, and maintaining processes, but they also commonly co-occur (upwards of 60%). Current PTSD and depression treatments typically focus on their respective disorders rather than on common processes that maintain psychopathology; and, importantly, they do not explicitly target positive adaptive processes associated with resilience. Decades of experimental studies, prospective studies, and psychotherapy trials have identified interconnected maladaptive and adaptive processes associated with persistent psychopathology after stressful, destabilizing events. These maladaptive processes include: 1) unproductive event processing; 2) avoidance; and 3) reward sensitivity and processing deficits. These processes prolong negative mood, interfere with adaptive coping and processing of emotional material, and increase sensitivity to future stressful life events. PATH (Positive Processes and Transition to Health) directly targets these maladaptive processes while also teaching parallel adaptive skills (constructive processing, approach, and positive emotion processing and reward seeking). Six, 90-min sessions target individuals who have experienced a destabilizing life event and have persistent stressor-related symptoms. PATH utilizes life event processing (revisiting, meaning making), focusing repeatedly on an identified destabilizing life event, positive life events, and future events as a framework to identify maladaptive processes and teach constructive processing skills. PATH has the potential to reduce dropout, improve treatment engagement and outcomes, identify potential treatment mechanisms, and ultimately reduce the costly human and economic burden of stressor-related psychopathology.

For the open trial's "Go" to be achieved and to proceed to the R33, two criteria must be met. The first is that at least 2 of the 3 primary targets must change via PATH. A moderate effect size (d = 0.60) was chosen to reflect evidence of clinically meaningful target engagement (see Gold et al., 2017), in line with NIMH guidelines for a preliminary signal of target engagement/efficacy in intervention trials. Second, at least one of the secondary measures must show a moderate effect (d = 0.50) from pre- to post-treatment. The investigators included measures of each of the targets, as they are conceptualized as interrelated parts of a "stuck" system. For "Go" to an R01 after the R33, in addition to target engagement, primary outcomes of PTSD and depression must show clinically meaningful gains (e.g., Barth et al., 2016; Cusak et al., 2016).

In the R33 phase, if the investigators achieve the "Go" criteria, the investigators will conduct a randomized controlled trial comparing PATH to PMR. PMR is a commonly used control condition that is rated as credible and helpful by patients. PMR will consist of six 60-90 minute sessions, focusing on stress management.

ELIGIBILITY:
Inclusion Criteria:

* Destabilizing life event involving profound loss or threat, with a minimum duration of 12 weeks since the event, but occurred within the last 5 years.
* Between the ages of 18 and 65.
* Elevated target: Scores of at least moderate (1 or higher) on at least 2 of the 3 target mechanisms: re- experiencing or ruminative processing of the destabilizing event (PSS-I items: 1, 2, 3, 4 or QIDS-C item 11), avoidance (PSS-I items 6, 7, 8), or reward deficits (PSS-I items 12, 13, or QIDS-C item 13).

Exclusion Criteria:

* Current diagnosis of schizophrenia, delusional disorder, or organic mental disorder as defined by DSM-5.
* Current diagnosis of bipolar disorder, depression with psychotic features, or depression severe enough to require immediate psychiatric treatment (i.e., serious suicide risk with intent and plan).
* Severe self-injurious behavior or suicide attempt within the previous three months.
* Unwilling or unable to discontinue current cognitive behavioral psychotherapy.
* No clear memory of the destabilizing event or event occurred before age 3.
* Unstable dose of psychotropic medications in prior 3 months.
* Ongoing intimate relationship with the perpetrator (in assault related event).
* Current diagnosis of a substance use disorder (DSM-5).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Affective Updating Task | Change from baseline score at 6 weeks (immediately post treatment)
  Measure updating of affective information in working memory
Idiographic Behavioral Approach Task | Change from baseline score at 6 weeks (immediately post treatment)
  Use in vivo confrontation with feared or avoided stimuli measuring avoidance behavior
Probabilistic Reward Task | Change from baseline score at 6 weeks (immediately post treatment)
  Assesses reward responsivity

SECONDARY OUTCOMES:
Posttraumatic Cognitions Inventory | Change from baseline score at 6 weeks (immediately post treatment)
  Self-report of negative, overgeneralized stressor-related thoughts
Behavioral Activation for Depression Scale | Change from baseline score at 6 weeks (immediately post treatment)
  Self-report of approach and avoidance in cognitive and behavioral domains (not specific to depression)
Snaith-Hamilton Pleasure Scale | Change from baseline score at 6 weeks (immediately post treatment)
  Self-report measuring the capacity to experience pleasure

CONTACTS AND LOCATIONS:
Overall Officials: Norah Feeny, PhD, Principal Investigator — Case Western Reserve University
Locations (3):
- United States (3):
  - University of Delaware, Newark, Delaware
  - Case Western Reserve University, Cleveland, Ohio
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-03-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT06093906/ICF_000.pdf